CLINICAL TRIAL: NCT03326804
Title: A Prospective, Non-randomized, Consecutive Series, Multicentre, Observational Study to Evaluate the Clinical Outcome of ceramic-on- Ceramic Hip Resurfacing Arthroplasty Using the Ceramic, Non-porous, Non-cemented H1 Hip Resurfacing Arthroplasty
Brief Title: H1 Hip Resurfacing Arthroplasty
Acronym: H1HRA
Status: Active, not recruiting | Type: Observational
Sponsor: Embody Orthopaedic Limited (Industry)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 213102
Record Dates: First submitted 2017-10-15; First posted 2017-10-31 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Hip Osteoarthritis; Hip Necrosis; Hip Dysplasia
Keywords: Hip Resurfacing Arthroplasty; Ceramic; Cementless; H1
MeSH Terms: conditions — Osteoarthritis, Hip; Hip Dislocation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 5 samples of 2ml of Blood stored in EDTA tubes will be taken and analysed for metal ion levels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1 - Safety: Cohort 1 will consist of the first 20 participants recruited into the study for H1 Hip Resurfacing Arthroplasty. These patients will receive additional CT scans preoperatively and then post-operatively at these time points: immediately postoperatively (2days), at 6 weeks, 3 months, 6 months, 1 year and 2 years. They will have metal-ion measurements for safety analysis. Blood samples will be taken preoperatively and postoperatively at 3 months, 6 months, 1 year and 2 years.
  A safety analysis of Cohort 1 will be performed at the 6 week, 3 month and 6 month post-operative stage by independent assessors. Yearly clinical evaluations will be performed until 10 years, and radiographs at 3,5,10 years. If the investigation supports the safety of the implant, the study will proceed with recruitment into Cohort 2.
  Interventions: Device: H1 Hip Resurfacing Arthroplasty
- Cohort 2 - Efficacy: Cohort 2 will consist of the remaining target size population of 230 patients for H1 Hip Resurfacing Arthroplasty. They will undergo the same intervention as previously described for Cohort 1, but will not undergo metal-ion testing and reduced frequency CT-scans.
  Interventions: Device: H1 Hip Resurfacing Arthroplasty

INTERVENTIONS:
Device: H1 Hip Resurfacing Arthroplasty — A non-porous non-cemented ceramic-on-ceramic hip resurfacing arthroplasty device

SUMMARY:
This is a prospective, non-randomized, consecutive series, multicentre, observational study to evaluate the clinical outcome of ceramic-on- ceramic hip resurfacing arthroplasty using the ceramic, non-porous, non-cemented H1 Hip Resurfacing Arthroplasty. It includes a safety study followed by an efficacy study. Patients will be followed up for 10-years postoperatively.

The primary aim is to confirm the safety of the H1 hip resurfacing prosthesis by demonstrating non-inferiority of the H1 device in terms of survivorship.

The secondary is to evaluate superiority of the ceramic-on-ceramic H1 hip resurfacing prosthesis compared to Metal-on-Metal (MoM) hip resurfacing in terms of absence of metal ion release.The primary end point is revision for any reason.

DETAILED DESCRIPTION:
Investigation type: Premarket study to receive a CE marking, followed by post-marketing surveillance follow-up.

Investigation design: Multi-centre, prospective, non-randomized, observational study

Investigation objectives:

The primary objective is to confirm the safety and efficacy of the H1 hip resurfacing prosthesis by demonstrating non-inferiority of the cumulative percent success in subjects implanted with the H1 hip resurfacing compared to a literature reference rate of the Birmingham hip resurfacing (BHR).

The secondary objective is to demonstrate superiority of the ceramic-on-ceramic H1 hip resurfacing prosthesis with its metal-free articulation compared to MoM hip resurfacing in the absence of metal ion release. Additional goals are to demonstrate non-inferiority of the ceramic-on-ceramic H1 hip resurfacing prosthesis compared to hip resurfacing with regard to patient reported outcome measures, objective clinical and functional outcomes, and radiological assessment.

The primary endpoint is revision for any reason

Secondary endpoints:

* Complication rate (adverse events and revisions)
* Toxicology (blood metal ion measurements)
* CT assessment (Implant migration)
* Patient Reported Outcome Measures (PROMs)
* Objective clinical and functional outcomes (Harris Hip Score, Gait Analysis)
* Radiological assessment (implant orientation, osseointegration)

Background Information

Total Hip Arthroplasty (THA) is one of the most successful surgical interventions. Replacement of an arthritic hip joint provides significant pain relief and improvement of hip function and mobility. Patients, even elderly people, are more active, have a better quality of life, less comorbidities and a longer life expectancy. The World Health Organisation (WHO) has declared THA the second best intervention, only preceded by cataract surgery, regarding cost effectiveness and quality of outcome. In patients older than 70 years, the overall survivorship of THA is more than 90% at 10 years and the best clinical results are obtained for THA as a treatment for osteoarthritis (OA). In this patient population, THA can thus be considered a lifelong solution. However, both survivorship and clinical results are much worse in young and active people. The reasons for this worse outcome are multiple. First of all, younger people usually have a more active lifestyle regarding work and sports. Secondly, the hip disorders leading to THA in a younger patient population are more difficult to treat. Congenital hip dysplasia is frequently associated with gross hip deformities, as may be the case in secondary traumatic OA. Bone stock may be jeopardised in cases of avascular necrosis of the femoral head (AVN) and rheumatoid arthritis (RA). Thirdly, a faster bone metabolism may play a role, but this remains to be elucidated.

Modern hip resurfacing arthroplasty (HRA) was introduced to address the inferior survivorship and unsatisfactory clinical results with THA in young and active patients. The anatomical reconstruction of the joint has the potential to provide a better function and higher activity levels compared to THA. Hip resurfacings are inherently higher performing than total hip replacements because they preserve the flexibility of native femoral head and neck. Metal-on-Metal (MoM) hip resurfacings have been shown to be safe and effective in many patients. These patients have superior clinical function over patients with total hip replacements, with little or no wear at the bearing surface in comparison to hard on soft bearings. The two most serious complications following hip surgery are death and infection. Both of these are substantially rarer after hip resurfacing when compared to patients with a cemented total hip arthroplasty, which is often presented as the gold standard of hip replacement. However, patients with poorly positioned hip resurfacing implants, poorly designed implants and smaller sizes especially in females have reported progressive pain leading to early revision. This pain is commonly caused by one of two problems: either metal ion particles generated by excessive wear associated with adverse soft tissue reactions to metal debris or soft tissue impingement on the hard metal edges of the components. Despite these two problems, hip registries continue to show superior survivorship of hip resurfacing using a well-designed device in young and active males when compared to total hip arthroplasty.

Higher metal ion levels have been found in whole blood, serum and urine of patients with MoM hip arthroplasties (THA and HRA) compared to preoperative values, and to THA with other bearing surfaces (metal-on-polyethylene, ceramic-on-polyethylene, ceramic-on-ceramic). Although MoM hip arthroplasty has been shown to produce less volumetric wear compared to metal-on-polyethylene, the wear debris consists of more numerous, small, nanometre size particles, which are ingested by macrophages. Contrary to polyethylene, metal particles and ions are not chemically inert but may have directly toxic, biological effects and may elicit hypersensitivity reactions in addition to the macrophage-driven, innate, foreign-body immune responses to particulate debris of any material. Consequently, concerns have been raised about the physiological consequences of metal release from MoM hip prostheses into the peri- prosthetic tissue and systemic circulation.

By exchanging the metal material of the bearing with BIOLOX®delta ceramic, a better wearing and more inert material, the positive clinical performance aspects of MoM hip resurfacings are retained, while the main cause of early revision is removed. The anatomic shape of the contours of the devices may go some way to reducing the pain caused by soft tissue erosion, Thus, the H1 ceramic-on-ceramic hip resurfacing could be used for wider indications than the currently restricted group of large men. Patients with smaller head sizes, females and patients with metal sensitivity may all be candidates, enabling them the option to have a more conservative operation if appropriate.

The H1 hip resurfacing design is innovative both in its anatomical shape and in the bearing couple materials as there is currently no all-ceramic bearing hip resurfacing implant in clinical use. Ceramic-on-ceramic THA has a proven track record with excellent survivorship results in the arthroplasty registries as well as low complication rates and good functional results from large clinical series. The materials have been thoroughly tested regarding biocompatibility, biomechanical and tribological characteristics, and have been used in over one million clinical cases over the last 11 years, confirming safety of the material. However, a mono-block ceramic acetabular component without a metal shell such as the H1 hip has not yet been used clinically. The concept requires investigation before it can be CE marked and marketed in Europe.

The anatomical contoured edge of both the cup and the head reduces the incidence of psoas impingement. The iliopsoas tendon is stretched over the femoral head when the hip is extended. In the normal hip, the tendon runs over the front edge of the acetabulum, and femoral head, which it uses as a fulcrum giving some leverage advantage as the muscle contracts to lift the leg up when bringing the leg up into the bath or into a high car for instance. When the femoral head is resurfaced, the tendon has to rub over the hard edge of the resurfacing device. Until now, femoral resurfacing devices have had a symmetric rim, which tends to extend beyond the normal limits of a femoral head, particularly in female hips. This overhang can cause painful abrasion of the tendon. Most acetabular components are also symmetric in shape, unlike the natural acetabular rim contour, which has a recess where the tendon runs. The rim of the acetabular shell can also be a cause of tendon irritation.

BIOLOX®delta is a zirconia toughened alumina (ZTA). Along with alumina (Al) and zirconia (Zr), this material also contains traces of chromium (Cr), strontium (Sr) and very low amounts of yttrium (Y). This ceramic has an 11-year history of worldwide use in hip arthroplasty, with an excellent track record. Ceramic-on-ceramic bearings consist of the hardest material with the lowest wear rate of all bearing couples used in hip arthroplasty. The very low volume of inert ceramic nanoparticles and the absence of elevated Cobalt (Co) and Cr ion levels in the bloodstream virtually abolishes the risk of adverse local tissue reactions (ALTR), allergic reactions and systemic cobalt toxicity which can complicate some MoM Hip replacements. BIOLOX®delta contains very small amounts of Cr, but Cr release from the material remains below the detection limit in the blood. Strontium ions are found in the blood of control patients without any implant and remain at similar background level in patients with BIOLOX®delta ceramic implants, Yttrium ions are not detected.

BIOLOX®delta is a zirconia-toughened alumina ceramic with increased fracture strengths. The use of BIOLOX®delta has virtually eliminated the already low fracture risk of the older ceramic implants. The fracture risk in the arthroplasty registries and as assessed by the manufacturer CeramTec is now estimated at < 0.001%.

Besides a significantly lower risk of mortality with hip resurfacing compared to conventional cemented total hip arthroplasty (THA), the use of BIOLOX®delta ceramic on ceramic bearings further reduces the risk of the most devastating complication associated with THA, i.e. periprosthetic infection . Because of a significant reduction in biofilm formation and adherence to ceramic surfaces (69%) compared to metal (92%) and highly cross-linked polyethylene (HXL PE) (100%), the risk of periprosthetic infection is significantly reduced, to <0.5% at 10 years compared to >1% with polyethylene bearings including HXL PE.

The uncemented fixation of the H1 hip resurfacing is not novel. The porous ingrowth coating of plasma sprayed titanium and hydroxyapatite has been applied by a leading implant coating specialist (Medicoat AG, Mägenwil, Switzerland). Acetabular cups using these coatings are now standard products with more than 15 years of experience. Several metal-on-metal hip resurfacing designs for non-cemented use, have successfully been implanted in large series of patients. Ti ions may be released as part of the bone ingrowth process of the non-cemented hip of knee prosthesis, but Ti_ions from Titaniumdioxyde (TiO2) coatings or Titanium-aluminum-vanadium (TiAlV) hip or knee arthroplasty components are not associated with toxic, teratogenic or carcinogenic reactions.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires primary hip arthroplasty due to degenerative joint disease (primary osteoarthritis, posttraumatic osteoarthritis, avascular necrosis, developmental hip dysplasia)
* Patient is eligible for hip resurfacing arthroplasty: i.e. has sufficient bone stock at the level of the femoral head (<1/3 necrosis of the head) and neck (not osteopenic/porotic, see exclusion criteria)
* Patient is between 18 and 70 years old
* Patient willing to comply with study requirements
* Patient is legally entitled and able to consent, agrees to consent to and to follow the study visit schedule (as defined in the study protocol and informed consent form), by signing the informed consent form approved by the Ethics Committee.
* Patient plans to be available through ten (10) years postoperative follow-up
* Patient is able to understand the native language of the country of the trial centre

Exclusion Criteria:

* Patient has a BMI greater than 40
* Patient suffers from an active inflammatory joint disorder
* Patient has an active infection or sepsis (treated or untreated)
* Patient has insufficient bone stock at the hip (>1/3 necrosis of the femoral head) or in general as in severe osteopenia or osteoporosis (Tscore < -2.5 as measured with BMD)
* At the time of enrolment, patient has one or more of the following arthroplasties that have been
* Implanted less than 6 months before the current hip arthroplasty:
* Contralateral primary total hip arthroplasty or hip resurfacing arthroplasty
* Ipsilateral or contralateral primary total knee or unicondylar knee arthroplasty
* Patient takes medications which potentially affect the bone such as corticosteroids and antimitotic medications.
* Patient has a condition that may interfere with the hip arthroplasty survival or outcome (i.e. Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease)
* Patient has a known alcohol or drug abuse
* Patient has an immunosuppressive disorder
* Patient has a malignant tumour, metastatic, or neoplastic disease
* Patient has severe comorbidities or a limited life expectancy
* Patient lacks capacity to consent
* Patient has an emotional or neurological condition that would pre-empt his/her ability or willingness to participate in the study
* Patient is not willing or able to sign an informed consent form
* Patient pregnant or breast feeding
* Patient is not able or willing to come to follow-up visits
* In addition, the following exclusion criteria are applied to the 20 patients (Cohort 1 and Cohort 1.1) in the safety study in whom metal ion measurements will be performed, since those conditions may be associated with elevated metal ion levels and could complicate the interpretation of the metal ion results:
* Patients who already received another joint replacement, hip, knee, shoulder, ankle.
* Workers in the paint, diamond, leather or other industries producing Co or Cr dust.
* Patients taking medication, vitamins or food supplements containing Co or Cr and not able or willing to discontinue those.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Indications for use of the H1 HRA in this investigation will be patients with end-stage hip disease who are candidates for primary hip arthroplasty using either a metal-on-metal hip resurfacing or a ceramic-on- ceramic THR. Typically they will be younger (<70 years) and active males and females with end-stage hip osteoarthritis, avascular necrosis of the femoral head, post-traumatic osteoarthritis or developmental dysplasia of the hip (DDH).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-09-26 (Actual); Primary Completion 2032-09-25 (Estimated); Study Completion 2033-03-25 (Estimated)

PRIMARY OUTCOMES:
Oxford Hip Score | 10 years
  Hip Specific Patient Reported Outcome Measure (PROM)
EQ-5D Health-Related Quality of Life Questionnaire | 10 years
  Generic Patient Reported Outcome Measure (PROM)

SECONDARY OUTCOMES:
Complication Rate | 10 years
  Adverse Events and revisions
Clinical objective outcome measures | 10 years
  Harris Hip Score
Acetabular Implant orientation | 10 years
  Evaluation of AP and Lateral Hip Radiographs, measured in degrees
Femoral Implant orientation | 10 years
  Evaluation of AP and Lateral Hip Radiographs, measured in degrees
Low-dose CT | Up till 2 years
  CT to evaluate component migration and bone ingrowth (Safety study - Cohort 1 - 20 patients)
Metal ion measurements | Up till 2 years
  Concentration of metal ions in patient's blood (Safety study - Cohort 1 - 20 patients)

CONTACTS AND LOCATIONS:
Overall Officials: Justin P Cobb, FRCS, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Charing Cross Hospital, London
  - Kind Edward VII's Hospital, London

IPD SHARING:
Plan to Share IPD: No